CLINICAL TRIAL: NCT06892652
Title: Feasibility and Effects of Comprehensive Management for Terminal Heart Failure (COMFORT-HF) Program: A Pilot Randomized Controlled Trial
Brief Title: Comprehensive Management for Terminal Heart Failure Program:
Acronym: COMFORT-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202408115RINA
Record Dates: First submitted 2025-03-10; First posted 2025-03-25 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
Keywords: palliative care; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supportive care (Experimental): supportive care
  Interventions: Other: Supportive care measures
- Control (No Intervention): usual care

INTERVENTIONS:
Other: Supportive care measures — shared decision making with patients and families to receive specialist palliative care
  Arms: supportive care

SUMMARY:
Advanced heart failure presents with various symptoms, including pain, dyspnea, functional decline, reduced quality of life, and physiological deterioration, which can ultimately lead to spiritual distress. The functional losses experienced by patients-encompassing physical, social, and mental aspects-place a significant burden on caregivers, impacting their physical, mental, and spiritual well-being. This burden is further intensified by the stress of making major medical decisions, highlighting the need for palliative care that extends beyond the patient. Addressing how to holistically support both patients and caregivers is a key focus of palliative care.

Studies have shown that integrating palliative care with heart failure treatment significantly improves patients' quality of life, as well as their comfort and dignity at the end of life. Evidence from multiple studies demonstrates the benefits of palliative care for heart failure patients, including enhanced quality of life, reduced emergency department visits and hospitalizations, and increased participation in advance care planning discussions. Consequently, national guidelines in several countries, including the United States and Europe, recommend the early integration of specialist palliative care for heart failure patients. However, the optimal timing for intervention by palliative care specialists remains undetermined.

This study aims to develop and assess the feasibility and effectiveness of the Comprehensive Management for Terminal Heart Failure (COMFORT-HF) program. Participants will be randomly assigned to either the experimental group, which will receive the COMFORT-HF model, or the control group, which will receive usual care. The implementation of the COMFORT-HF model involves heart failure case managers conducting screenings to identify patients for referral to a specialist palliative care team. Once the shared decision-making process is initiated and both the patient and the primary heart failure care team agree, palliative care specialists and shared care nurses will collaborate with the heart failure team to provide comprehensive, coordinated care, including regular visits.

The study aim to validate that the COMFORT-HF model produces positive outcomes for patients with advanced heart failure, making it a promising approach for broader implementation and promotion.

ELIGIBILITY:
Inclusion Criteria:

1. Congestive heart failure at stage C or D
2. Age ≥ 18 years
3. Able to communicate in Chinese or Taiwanese

Exclusion Criteria:

1. Pregnant women
2. Patients who have previously received palliative care services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | days 0, months 6, months 12
  The EQ-5D-5L is a standardized instrument for measuring generic health-related quality of life. It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity: no problems, slight problems, moderate problems, severe problems, and extreme problems.
  Scoring Range: The EQ-5D-5L utility score ranges from -0.594 to 1, where 1 represents full health, 0 represents death, and negative values represent health states worse than death.
  Interpretation: Higher scores indicate better health-related quality of life.

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire | Day 0, months 6, months 12
  The KCCQ is a disease-specific instrument designed to assess health status in heart failure patients. It includes multiple domains: physical limitation, symptom frequency, symptom burden, social limitation, and quality of life. The questionnaire generates an overall Total Summary Score (TSS).
  Scoring Range:
  Each domain score ranges from 0 to 100. The Total Summary Score (TSS) ranges from 0 to 100. Interpretation: Higher scores indicate better health status, fewer symptoms, and improved quality of life. A lower score represents worse symptoms and greater functional impairment.
Quality of Dying Evaluation Form in the Hospice and Palliative Care Unit at National Taiwan University Hospital | During the intervention, If patient passed away
  This is a validated tool specifically designed to assess the quality of dying in terminally ill patients receiving hospice and palliative care. It evaluates multiple aspects, including symptom control, comfort, dignity, emotional support, and communication.
  score ranging from 0 to 15 to summarize the extent to which the death was considered good. Interpretation: Higher scores indicate better quality of dying (e.g., better symptom relief, patient dignity, and family satisfaction), while lower scores suggest greater suffering or unmet needs.
Spiritual well-being scale | Day 0, months 6, months 12
  The SWBS is a self-report questionnaire assessing two dimensions of spiritual well-being: Religious Well-Being (RWB) (connection to a higher power) and Existential Well-Being (EWB) (sense of life meaning and satisfaction). It consists of 20 items.
  Scoring Range:
  Each item is scored on a 6-point Likert scale (1 = strongly disagree, 6 = strongly agree).
  The total score ranges from 20 to 120. The Religious Well-Being subscale ranges from 10 to 60, and the Existential Well-Being subscale also ranges from 10 to 60.
  Interpretation: Higher scores indicate greater spiritual well-being, while lower scores suggest spiritual distress or dissatisfaction.

IPD SHARING:
Plan to Share IPD: Yes
The data was available under reasonable request to responsible authors
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available after acceptance of the submission to journal
Access Criteria: reasonable request to corresponding author